CLINICAL TRIAL: NCT02563652
Title: Can Biomarkers Aid in the Prediction of Postoperative Pain and Circulatory Instability After Major Abdominal Surgery? A Prospective Observational Study
Brief Title: Can Biomarkers Aid in the Prediction of Postoperative Pain and Circulatory Instability After Major Abdominal Surgery?
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: University of Parma (Other); Study in Multidisciplinary Pain Research Group, Italy (Unknown); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/641
Record Dates: First submitted 2015-09-08; First posted 2015-09-30 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Abdomen/surgery; Biological markers; Length of stay; Postoperative care; Anesthesia recovery period; Prognosis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood, serum, plasma and urine will be stored in cryotubes at -81 degrees celcius for later analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major abdominal surgery: Patients undergoing major abdominal surgery (laparotomy). Surgical procedures considered for inclusion include, but are not restricted to, procedures such as gastrectomy, pancreatic surgery, liver resection, open prostatectomy, colonic surgery, radical cystectomy with ileal conduit, open nephrectomy and vascular abdominal aortic surgery.

SUMMARY:
Patients undergoing major surgery are exposed to extensive damage of tissues, which induces widespread activation of the inflammatory system, called 'systemic inflammatory response syndrome' (SIRS).This activation of the inflammatory system may induce instability of the heart and respiration in the postoperative period. The degree of physiologic response to postoperative SIRS as well as the degree of postoperative pain differ between patients. Therefore, patients undergoing anesthesia and major surgery are treated in a 'post anesthesia care unit' (PACU) after end of surgery.Admittance to a PACU is expensive. The time patients need to stay in a PACU after major surgery has not been extensively studied, and more appropriate tools for prediction of length of stay are needed.

The main aim of this study is to assess whether clinical observations, inflammatory biomarkers or genetic markers may aid in the prediction of physiological instability and/or pain after major surgery. Such predictors would help clinicians planning the length of PACU-stays.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major abdominal surgery (e.g. Whipple's operation, liver resection, abdominoperineal resection, vascular abdominal surgery etc.)
* Scheduled for PACU stay first 24 hours

Exclusion Criteria:

* Pregnancy
* Jehovah's witness
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for major abdominal surgery in St Olavs Hospital, Trondheim, Norway
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Time to established circulatory stability for > 2 hours [Time to event outcome] | 48 hours
  Circulatory stability will be assessed by applying a multi-state statistical model, where any state changes are measured at an hourly basis. The model will include variables reflecting the circulatory state of the patient, including heart rate, systolic blood pressure (or MAP) and lactate, which will be assessed together with the measures needed to maintain them, such as the amount of fluid given (ml per hour) and the extent of vasopressor (i.e. norepinephrine). The main outcome variable will be the time needed to reach the state of 'stable without intervention for more than two hours. To be classified in this state, the systolic blood pressure must be > 100 mmHg, the heart rate between 40 and 110, the patient must be off vasopressor and has a fluid requirement of less than 250 ml/hour.
Time to reaching a state of no or mild pain problem for > 2 hours [Time to event outcome] | 48 hours
  This outcome will be reached when the patient has a numeric rating score (NRS) with respect to pain of < 4 and the opioid consumption is less than 5 mg morphine equivalents per hour.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Solligård, phd md, Study Director — St. Olavs Hospital
Locations (2):
- University of Parma, Parma, Italy
- St Olavs Hospital, Trondheim, Norway